CLINICAL TRIAL: NCT01079299
Title: Intermittent, Gradient, Pneumatic Compression Plus Standard Compression for Hard-To-Heal Venous Ulcers in Subjects With Secondary Lymphedema and Chronic Venous Insufficiency
Brief Title: Effect of Intermittent Pneumatic Compression on Ulcer Healing in Subjects With Secondary Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calvary Hospital, Bronx, NY (Other)
Collaborators: RTS Family Foundation (Unknown); New York State Department of Health (Other Government)
Responsible Party: Oscar M. Alvarez, PhD / Principal Investigator, Center for curative and Palliative Wound Care, Calvary Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-VU-0308
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2012-02-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2010-08

CONDITIONS: Lymphedema
Keywords: venous ulcer; secondary lymphedema; chronic lower leg ulceration
MeSH Terms: conditions — Lymphedema; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPC plus standard compression (Experimental)
  Interventions: Device: Intermittent, gradient, pneumatic compression device
- Standard compression alone (Active Comparator)
  Interventions: Device: Intermittent, gradient, pneumatic compression device

INTERVENTIONS:
Device: Intermittent, gradient, pneumatic compression device — lymphedema pump provides external compression in a segmental,gradient fashion
  Other Names: Bio 4000 (Bio Compression Inc, Moonachie,NJ)

SUMMARY:
This is a randomized, controlled, parallel group, open label, clinical trial to evaluate the effectiveness of intermittent, gradient, pneumatic compression (IPC)on the healing of venous ulcers in subjects diagnosed with chronic secondary lymphedema. Time to complete healing, healing rates, edema, wound pain, granulation tissue, and wound exudate (type and amount) will be compared between the IPC-treated group (IPC plus standard compression)and control (standard compression alone).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with secondary lymphedema
* Presence of a venous ulcer that has not healed in more than 6 months
* Localized wound pain greater than 3 with VAS
* Ulcer must be on lower leg (below knee)
* Ulcer must be of venous etiology
* CVI proven by duplex studies
* Subject must have adequate arterial blood flow (ABI > 0.70)
* Subject must be able to tolerate compression bandages
* Subject must be ambulatory
* Capable of understanding consent process

Exclusion Criteria:

* Wound infection
* Ulcer of non-venous etiology
* Ulcer on toes or plantar surface of the foot
* Subject taking any medication that in the opinion of the investigator affects wound healing
* Alcohol or drug abuse
* Active deep venous thrombosis (DVT)
* Subject has a cancer diagnosis
* Diabetic with hemoglobin A1C>12
* Arterial insufficiency ABI<0.70
* Subject is not capable of walking (wheelchair-bound or bed-bound)
* Subject currently enrolled in another clinical trial
* Moderate to severe congestive heart failure

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-12; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Calvary Hospital, Center for Curative and Palliative Wound Care, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 52 subjects were treated, IPC n=27, Control n=25
Period: Overall Study
Arm/Group | IPC Plus Standard Compression | Standard Compression Alone
Started | 27 | 25
Completed | 27 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IPC Plus Standard Compression | Standard Compression Alone | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 16 | 12 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (5.6) | 59 (4.9) | 62 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Wound Closure at 9 Months
Description: Median number of days for complete healing in each treatment group
Time Frame: 9 months
Measure: Median (Standard Error); unit: median number of days for complete heali
Arm/Group | IPC Plus Standard Compression | Standard Compression Alone
Number analyzed (Participants) | 27 | 25
median number of days for complete heali | 141 (24) | 211 (29)

ADVERSE EVENTS:
Arm/Group | IPC Plus Standard Compression | Standard Compression Alone
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No